CLINICAL TRIAL: NCT06316973
Title: A Phase 1a, Randomized, Double-Blind, Placebo-Controlled, Single Center Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CS-1103 Following Single, Ascending Intravenous Dose Administration in Healthy Participants
Brief Title: A Clinical Study to Evaluate the Safety of CS-1103 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clear Scientific, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS-1103-01; U01DA053054 (NIH)
Record Dates: First submitted 2024-03-05; First posted 2024-03-19 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Substance Use Disorders; Methamphetamine Abuse; Methamphetamine Intoxication
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Single Center Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CS-1103 Following Single, Ascending Intravenous Dose Administration in Healthy Participants
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): 6 participants received a single dose of 2.7 mg/kg (2.5 mg/kg free acid) CS-1103 administered as solution for infusion by IV over 10 minutes.
  A diluted CS-1103 saline solution in an IV bag is used for drug administration.
  Interventions: Drug: CS-1103
- Cohort 2 (Experimental): 6 participants received single dose of 8.0 mg/kg (7.5 mg/kg free acid) CS-1103 administered as solution for infusion by IV over 10 minutes.
  A diluted CS-1103 saline solution in an IV bag is used for drug administration.
  Interventions: Drug: CS-1103
- Cohort 3 (Experimental): 6 participants received a single dose of 16.0 mg/kg (15.1 mg/kg free acid) CS-1103 administered as solution for infusion by IV over 10 minutes.
  A diluted CS-1103 saline solution in an IV bag is used for drug administration.
  Interventions: Drug: CS-1103
- Cohort 4 (Experimental): 6 participants received a single dose of 19.0 mg/kg (17.9 mg/kg free acid) CS-1103 administered as solution for infusion by IV over 10 minutes.
  A diluted CS-1103 saline solution in an IV bag is used for drug administration.
  Interventions: Drug: CS-1103
- Placebo (Placebo Comparator): 2 participants for each cohort were administered with placebo.
  Total administered volume of saline matched administered volume for the corresponding CS-1103 solution in each cohort.
  Interventions: Drug: Sterile Saline

INTERVENTIONS:
Drug: CS-1103 — CS-1103 for infusion
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: Sterile Saline — Sterile Saline for Injection
  Arms: Placebo

SUMMARY:
The purpose of this Phase 1a study is to evaluate safety, tolerability, and pharmacokinetics (PK) of single, ascending doses of CS-1103, administered by intravenous (IV) infusion in healthy participants.

ELIGIBILITY:
Major Inclusion Criteria:

1. Healthy male and/or female participants aged 18 to 55 years, inclusive.
2. A body mass index between 18.0 to 30.0 kg/m2, inclusive, and a minimum body weight of 50 kg.
3. Females must be of nonchildbearing potential.

Major Exclusion Criteria:

1. Estimated glomerular filtration rate <90 mL/min/1.73 m2
2. Any clinically significant abnormalities in rhythm, conduction or morphology of the resting ECG, and any clinically important abnormalities in the 12-lead ECG
3. Current smokers, or those who have smoked or used nicotine products (including nicotine patches) within 1 month prior to dose administration.
4. History of alcohol abuse or excessive intake of alcohol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Vince Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (2.5 mg/kg CS-1103 [Free Acid]): 6 participants received a single dose of 2.7 mg/kg (2.5 mg/kg free acid) CS-1103 administered as solution for infusion by IV over 10 minutes.
  A diluted CS-1103 saline solution in an IV bag is used for drug administration.
- Cohort 2 (7.5 mg/kg CS-1103 [Free Acid]): 6 participants received single dose of 8.0 mg/kg (7.5 mg/kg free acid) CS-1103 administered as solution for infusion by IV over 10 minutes.
  A diluted CS-1103 saline solution in an IV bag is used for drug administration.
- Cohort 3 (15.1 mg/kg CS-1103 [Free Acid]): 6 participants received a single dose of 16.0 mg/kg (15.1 mg/kg free acid) CS-1103 administered as solution for infusion by IV over 10 minutes.
  A diluted CS-1103 saline solution in an IV bag is used for drug administration.
- Cohort 4 (17.9 mg/kg CS-1103 [Free Acid]): 6 participants received a single dose of 19.0 mg/kg (17.9 mg/kg free acid) CS-1103 administered as solution for infusion by IV over 10 minutes.
  A diluted CS-1103 saline solution in an IV bag is used for drug administration.
Period: Overall Study
Arm/Group | Cohort 1 (2.5 mg/kg CS-1103 [Free Acid]) | Cohort 2 (7.5 mg/kg CS-1103 [Free Acid]) | Cohort 3 (15.1 mg/kg CS-1103 [Free Acid]) | Cohort 4 (17.9 mg/kg CS-1103 [Free Acid]) | Placebo
Started | 6 | 6 | 6 | 6 | 8
Completed | 6 | 6 | 6 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (2.5 mg/kg CS-1103 [Free Acid]) | Cohort 2 (7.5 mg/kg CS-1103 [Free Acid]) | Cohort 3 (15.1 mg/kg CS-1103 [Free Acid]) | Cohort 4 (17.9 mg/kg CS-1103 [Free Acid]) | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (10.7) | 30.3 (8.3) | 39.5 (9.0) | 38.5 (7.9) | 36.3 (10.4) | 34.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 0 | 0 | 4
  Male | 6 | 5 | 3 | 6 | 8 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2 | 0 | 4
  Not Hispanic or Latino | 6 | 4 | 6 | 4 | 8 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 5 | 2 | 6 | 18
  White | 4 | 2 | 1 | 4 | 2 | 13
  More than one race | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.815 (2.479) | 24.728 (3.451) | 24.528 (2.731) | 25.975 (2.602) | 26.161 (2.308) | 25.487 (2.624)
Weight [Mean (Standard Deviation); unit: kg] | 83.30 (11.81) | 72.97 (8.30) | 68.32 (6.93) | 76.20 (9.27) | 79.44 (6.77) | 76.26 (9.60)
Height [Mean (Standard Deviation); unit: cm] | 179.23 (6.59) | 170.80 (10.11) | 166.97 (6.65) | 171.12 (5.98) | 174.63 (5.42) | 172.68 (7.73)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs)
Description: Treatment-emergent adverse events assessed through physical examinations, vital signs (blood pressure, pulse rate, respiratory rate, oxygen saturation, and body temperature), electrocardiograms (digital 12-lead electrocardiograms (ECGs). Any correlation between CS-1103 plasma concentrations and changes in QT intervals will be noted), and laboratory parameters (clinical chemistry, hematology, coagulation, and urinalysis).
Time Frame: 3 days plus 8 days for follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (2.5 mg/kg CS-1103 [Free Acid]) | Cohort 2 (7.5 mg/kg CS-1103 [Free Acid]) | Cohort 3 (15.1 mg/kg CS-1103 [Free Acid]) | Cohort 4 (17.9 mg/kg CS-1103 [Free Acid]) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants
  TEAEs | 1 | 1 | 2 | 4 | 0
  Related TEAEs | 0 | 0 | 1 | 4 | 0
  Serious TEAEs | 0 | 0 | 0 | 0 | 0
  TEAEs leading to study discontinuation | 0 | 0 | 0 | 0 | 0
  TEAEs leading to death | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants by Severity of AEs
Description: Severity of AEs was classified as mild, moderate, or severe (increasing severity).
  A subject experiencing multiple occurrences of an adverse event in a particular category was counted, at most, once for that category for each treatment.
Time Frame: 3 days plus 8 days for follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (2.5 mg/kg CS-1103 [Free Acid]) | Cohort 2 (7.5 mg/kg CS-1103 [Free Acid]) | Cohort 3 (15.1 mg/kg CS-1103 [Free Acid]) | Cohort 4 (17.9 mg/kg CS-1103 [Free Acid]) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants
  Mild | 1 | 1 | 2 | 4 | 0
  Moderate | 0 | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Plasma Pharmacokinetic (PK) Parameter: Cmax
Description: Maximum concentration, obtained directly from the observed concentration versus time data.
Time Frame: End-of-Infusion (EOI), 5, 10, 20, 30, 40 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 hr
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Cohort 1 (2.5 mg/kg CS-1103 [Free Acid]) | Cohort 2 (7.5 mg/kg CS-1103 [Free Acid]) | Cohort 3 (15.1 mg/kg CS-1103 [Free Acid]) | Cohort 4 (17.9 mg/kg CS-1103 [Free Acid])
Number analyzed (Participants) | 6 | 6 | 6 | 6
μg/mL | 20.78 (31.3) | 58.25 (17.7) | 156.9 (24.8) | 176.0 (17.9)

4. Secondary Outcome: Plasma PK Parameter: Tmax
Description: Time of maximum observed blood plasma concentration (Cmax) of CS-1103
Time Frame: End-of-Infusion (EOI), 5, 10, 20, 30, 40 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 hr
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 (2.5 mg/kg CS-1103 [Free Acid]) | Cohort 2 (7.5 mg/kg CS-1103 [Free Acid]) | Cohort 3 (15.1 mg/kg CS-1103 [Free Acid]) | Cohort 4 (17.9 mg/kg CS-1103 [Free Acid])
Number analyzed (Participants) | 6 | 5 | 6 | 5
hours | 0.235 [0.180 to 0.270] | 0.180 [0.180 to 0.330] | 0.180 [0.180 to 0.330] | 0.180 [0.180 to 0.250]

5. Secondary Outcome: Plasma PK Parameter: t1/2
Description: Terminal Elimination Half-life of CS-1103
Time Frame: End-of-Infusion (EOI), 5, 10, 20, 30, 40 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 hr
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Cohort 1 (2.5 mg/kg CS-1103 [Free Acid]) | Cohort 2 (7.5 mg/kg CS-1103 [Free Acid]) | Cohort 3 (15.1 mg/kg CS-1103 [Free Acid]) | Cohort 4 (17.9 mg/kg CS-1103 [Free Acid])
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 4.323 (26.4) | 4.118 (13.7) | 4.215 (17.4) | 4.558 (19.9)

6. Secondary Outcome: Plasma PK Parameter: CL
Description: Systemic Clearance of CS-1103
Time Frame: End-of-Infusion (EOI), 5, 10, 20, 30, 40 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 hr
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Cohort 1 (2.5 mg/kg CS-1103 [Free Acid]) | Cohort 2 (7.5 mg/kg CS-1103 [Free Acid]) | Cohort 3 (15.1 mg/kg CS-1103 [Free Acid]) | Cohort 4 (17.9 mg/kg CS-1103 [Free Acid])
Number analyzed (Participants) | 6 | 5 | 6 | 5
L/h | 0.04915 (24.2) | 0.04971 (16.1) | 0.04762 (20.6) | 0.05040 (17.3)

7. Secondary Outcome: Plasma PK Parameter: Vz
Description: Volume of Distribution of CS-1103
Time Frame: End-of-Infusion (EOI), 5, 10, 20, 30, 40 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 hr
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Cohort 1 (2.5 mg/kg CS-1103 [Free Acid]) | Cohort 2 (7.5 mg/kg CS-1103 [Free Acid]) | Cohort 3 (15.1 mg/kg CS-1103 [Free Acid]) | Cohort 4 (17.9 mg/kg CS-1103 [Free Acid])
Number analyzed (Participants) | 6 | 5 | 6 | 5
L | 0.3065 (15.0) | 0.2953 (7.8) | 0.2896 (12.0) | 0.3273 (24.0)

8. Secondary Outcome: Urine PK Parameter: Fe (0-last)
Description: Cumulative fraction of dose excreted in urine during the pooled collection intervals. Due to inherent error in measuring CS-1103 recovered in urine, the calculated recovery may exceed 100% of the dose.
Time Frame: Time intervals from 0-24 hours after IV administration of CS-1103
Measure: Mean (Standard Deviation); unit: percentage of dose administered
Arm/Group | Cohort 1 (2.5 mg/kg CS-1103 [Free Acid]) | Cohort 2 (7.5 mg/kg CS-1103 [Free Acid]) | Cohort 3 (15.1 mg/kg CS-1103 [Free Acid]) | Cohort 4 (17.9 mg/kg CS-1103 [Free Acid])
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage of dose administered | 91.58 (12.37) | 108.3 (4.227) | 101.0 (5.433) | 98.70 (9.129)

ADVERSE EVENTS:
Time Frame: 3 days plus 8 days for follow-up
Arm/Group | Cohort 1 (2.5 mg/kg CS-1103 [Free Acid]) | Cohort 2 (7.5 mg/kg CS-1103 [Free Acid]) | Cohort 3 (15.1 mg/kg CS-1103 [Free Acid]) | Cohort 4 (17.9 mg/kg CS-1103 [Free Acid]) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 2/6 | 4/6 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (2.5 mg/kg CS-1103 [Free Acid]) (N=6) | Cohort 2 (7.5 mg/kg CS-1103 [Free Acid]) (N=6) | Cohort 3 (15.1 mg/kg CS-1103 [Free Acid]) (N=6) | Cohort 4 (17.9 mg/kg CS-1103 [Free Acid]) (N=6) | Placebo (N=8)
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 1 | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT06316973/Prot_001.pdf
  • Statistical Analysis Plan (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT06316973/SAP_002.pdf
  • Informed Consent Form (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT06316973/ICF_000.pdf